CLINICAL TRIAL: NCT04606810
Title: Measuring the Impact of an Innovative Educational Intervention in Inflammatory Arthritis: a Natural Evolution of the Centre Hospitalier Universitaire (CHU) de Québec's Multidisciplinary Information Session
Brief Title: Measuring the Impact of an Innovative Educational Intervention in Inflammatory Arthritis
Acronym: I3A
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties at recruiting enough participants for this study
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: Canadian Rheumatology Association (Other); The Arthritis Society, Canada (Other); Laval University (Other); CISSS de Chaudière-Appalaches (Other Government); Clinique Rhumatologie/Physiatrie Centre du Québec, Trois-Rivières (Unknown); Centre de Rhumatologie de l'Est du Québec (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: MP-20-2015-2242
Record Dates: First submitted 2020-10-19; First posted 2020-10-28 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Rheumatoid Arthritis
Keywords: Patient therapeutic education; BioSecure questionnaire; Theory of planned behavior; Beliefs about medicines questionnaire
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: Participants in group 1 received the usual care plus the multidisciplinary educational intervention at baseline.
  Participants in group 2 first received usual care, and after 3 months were offered the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm1, Participants received the multidisciplinary educational intervention at baseline (Active Comparator): Participants in arm1 received the usual care plus the multidisciplinary educational intervention consisting of an educational DVD followed by a teleconference at baseline.
  Interventions: Other: multidisciplinary educational intervention
- Arm2, Participants in arm2 received the educational intervention after 3 months (Other): Participants in group 2 first received usual care, and after 3 months were offered the multidisciplinary educational intervention.
  Interventions: Other: multidisciplinary educational intervention

INTERVENTIONS:
Other: multidisciplinary educational intervention — At randomization, participants in arm 1 received the educational DVD with the instruction to review its contents within the next two weeks. Between 2 and 4 weeks after randomization, reinforcement teleconferences were done in small groups of 10 participants maximum per session with every participant who mentioned having watched the DVD. Each participant attended only to one teleconference. Usual care consisted in regular follow-up with the treating rheumatologist and possibility of asking questions of the rheumatology nurse by phone.

SUMMARY:
Self-management is critical for patients with chronic conditions such as rheumatoid arthritis. Such management requires that patients understand what to do to best manage their condition. This study will use a randomized controlled study design to evaluate the impact of a new educational intervention consisting of an educational digital video disc (DVD) and a self-management support session/teleconference with a multidisciplinary team of health care providers for patients (n=150) with active rheumatoid arthritis (RA) starting on or changing biologic agents. This study aims to test whether this intervention improves behavioural intentions, knowledge, and medication adherence three months post-intervention and whether acquired knowledge is retained six months after the intervention. This project will allow to quantify the impact of the educational intervention on patients' behavioural intentions in practical situations using an existing validated questionnaire called BioSecure. The impact of the educational intervention on disease-specific knowledge and on medication adherence will be evaluated using validated questionnaires.

DETAILED DESCRIPTION:
The primary objective of this study was to determine whether patients with active RA starting or changing biological agents demonstrate better self-care safety skills in practical situations using the BioSecure questionnaire three months after receiving a multidisciplinary educational intervention, as compared to patients who received usual care. The secondary objectives were to assess the impact of the educational intervention on behavioral intentions and beliefs and adherence to RA medications in patients receiving the intervention compared to usual care.

Trial design This was a pilot, unblinded, randomized study. Participants in group 1 received the usual care plus the multidisciplinary educational intervention at baseline. Participants in group 2 first received usual care, and after 3 months were offered the intervention. The patients' self-care safety skills was measured using the BioSecure questionnaire, and the behavioral intentions and beliefs with respect to medications was assessed using structured questionnaires at baseline, 3 and 6 months. With the participant authorization, data on RA medication adherence, i.e. biological agents and other non-biologic Disease-modifying anti-rheumatic drugs (nbDMARDs) was obtained for the 3 months preceding enrollment and up to 6 months afterwards using their pharmacy records.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years and had a diagnosis of RA,
* with active disease as per rheumatologist evaluation,
* having received a trial of two traditional nbDMARDs therapy, and
* who requires the addition or change of a biological agent

Exclusion Criteria:

* patient unable to consent,
* patient unable to answer questionnaires,
* patient unable to view a DVD at home
* patient unable to participate in a teleconference

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-10-07 (Actual)

PRIMARY OUTCOMES:
Change of knowledge on self-care safety skills | Change from baseline knowledge on self-care safety skills at 3 months.
  To measure the knowledge on self-care safety skills, the BioSecure questionnaire was used. This 55-item questionnaire measures the self-care safety skills of patients treated by biologic agent by the use of both knowledge and coping items. This questionnaire mainly contains true or false questions to assess patient's knowledge. Each good answer is given one point. The sum of points is then transformed into a percentage. A value of 100% represents a patient with perfect knowledge.

SECONDARY OUTCOMES:
Change of behavioral intention | Change of baseline behavioral intention at 6 months.
  According to published data on the Theory of Planned Behavior, a questionnaire to evaluate behavioral intention was developed, focussing on the appropriate or inappropriate intention to take an injection of a biologic agent while presenting symptoms of infection. It comprises 12 questions to be answered by the use of a 7-point Likert scale, from "Completely disagree" to "Completely agree". High values correspond to good attitude, norm, control or intention. There were 2 questions on attitude, 6 questions on perceived norms, 2 questions on perceived behavioral control, 1 question on intention, and 1 question on past behavior. Intention was dichotomized for analysis purpose, with values 1 to 3 considered as health-promoting intentions, while values 4 to 7 were health-damaging intentions.
Change of medication beliefs | Change of baseline medication beliefs at 6 months.
  For medication beliefs, the Belief about Medicines Questionnaire (BMQ) was adapted from the literature to RA medication. This questionnaire consists of 18 questions to evaluate the four sub-scales of the BMQ, ie specific-necessity (5 questions), specific-concern (5 questions), general-harm (4 questions), and general-overuse (4 questions), to be completed by selecting one item among five choices from "completely agree" to "completely disagree". The score of each subscale is the sum of its items, and thus has a maximum value of 25 or 20 points depending on its number of items. A high value corresponds to greater necessity, concern, harm or overuse.
Change of medication adherence | Change of medication adherence from 3 months before the study to 6 months
  Medication adherence was assessed using pharmacy records data. The proportion of adherence was calculated by dividing the quantity received by the quantity prescribed, separately for biologic agents and nbDMARDs, for each month starting 3 months before enrolment until 6 months after. For each time period (3 months before the study to baseline, baseline to 3 months, and 3 months to 6 months), the mean proportion of adherence per medication was then calculated taking the mean of all months included in each of the three periods. For each of these periods, the patient was considered to be adherent if the mean was equal to 100%. However, sensitivity analyses for adherence were also conducted using a threshold greater or equal to 80%, which is used in most clinical studies

IPD SHARING:
Plan to Share IPD: No